CLINICAL TRIAL: NCT06557642
Title: Investigating the Neuropsychological Effects of Nitrous Oxide
Brief Title: Nitrous Oxide and EMOtional Cognition
Acronym: NEMO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NEMO_Study
Record Dates: First submitted 2024-07-19; First posted 2024-08-16 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Depression
Keywords: Healthy Volunteers
MeSH Terms: conditions — Depression | interventions — Entonox; Air

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ENTONOX (50% nitrous oxide:50% oxygen) (Experimental): ENTONOX to be administered for 30 minutes.
  Interventions: Drug: Entonox
- Medical Air (Placebo Comparator): Medical Air to be administered for 30 minutes.
  Interventions: Drug: Medical Air

INTERVENTIONS:
Drug: Entonox — 30 minute inhalation using demand valve and mouthpiece
  Arms: ENTONOX (50% nitrous oxide:50% oxygen)
Drug: Medical Air — 30 minute inhalation using demand valve and mouthpiece
  Arms: Medical Air

SUMMARY:
The goal of this study is to uncover the underlying neuropsychological mechanisms of nitrous oxide, which may be relevant to its reported antidepressant effects. In particular, the study is designed to determine whether nitrous oxide changes the way in which healthy volunteers aged 18-40 years remember negative autobiographical memories.

The main question the study aims to answer is:

• Does nitrous oxide interfere with the emotional aspects of negative autobiographical memories?

Other neuropsychological effects will also be assessed (e.g., emotional processing, emotional memory, response inhibition, and cognitive flexibility).

Researchers will compare ENTONOX (50% nitrous oxide: 50% oxygen) with medical air.

Participants will:

* Attend three research visits (screening, inhalation, follow-up)
* Take part in a 30 minute inhalation session of ENTONOX or medical air
* Complete a series of cognitive tasks
* Finish a series of self-report questionnaires

DETAILED DESCRIPTION:
Questions regarding the mechanisms of nitrous oxide and its effects on the brain and behaviour in the context of its reported antidepressant effects remain largely unanswered. Thus, in the present study, the investigators aim to elucidate the more general effects that nitrous oxide might have on a series of neurocognitive processes which may be relevant to the treatment of depression. Namely, the study will investigate: 1) reconsolidation of autobiographical memories, 2) measures of emotional processing and emotional memory, 3) response inhibition, 4) cognitive flexibility and 5) sleep stages.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-40 years
* Good vision and hearing
* Willing and able to give informed consent
* Body mass index (BMI) within the range of 18-35kg/m2 (This is to ensure we exclude underweight individuals who might have more substantial reactions to the nitrous oxide).
* Sufficiently fluent in English to understand tasks
* Willing to avoid drinking any alcohol from 3 days prior to Visit One until the end of Visit Three
* Willing to avoid using recreational drugs for 3 months prior to Visit One and throughout the duration of the study

Exclusion Criteria:

* Receiving or seeking treatment for any mental health condition (covered in Structured Clinical Interview for the Diagnostic and Statistical Manual of Mental Disorders-5 (SCID) assessment in screening procedures)
* History of any mental health condition (covered in SCID assessment in screening procedures)
* Attention deficit hyperactivity disorder (ADHD) requiring treatment with stimulant or other centrally-acting drugs
* A positive drug test for any of the following: amphetamine, barbiturates, benzodiazepines, buprenorphine, cocaine, marijuana, methadone, methamphetamine, methylenedioxymethamphetamine (MDMA), morphine, methaqualone, opiates, phencyclidine, propoxyphene, tricyclic antidepressants, tramadol, ketamine, oxycodone, cotinine, 2-ethylidene-1,5-dimethyl-3,3-diphenylpyrrolidine (EDDP), fentanyl, synthetic marijuana, 6-mono-acetyl-morphine (6-MAM).
* Regularly drink 14 or more units of alcohol a week
* Any eye, throat or ear surgery or a medical procedure requiring intravenous injection or line into a vein in the last 6 months
* A head injury causing concussion or unconsciousness in the past 6 months
* A collapsed lung or lung surgery (e.g., pneumothorax)
* A history of cardiac arrhythmias
* Current injuries of the face or mouth (including ulcers or dental problems)
* Dental surgery in the past month
* Deep diving or scuba diving (which has a risk of decompression sickness) in past month
* Pregnancy / intention to become pregnant during the study
* Breastfeeding during the study
* Asthma, emphysema or any medical condition that affects the lungs or breathing
* Diagnosed vitamin B12 deficiency
* Any use of recreational drugs in the last three months
* Participation in any other drug study in the last three months
* Participation in any other study with the same tasks in the last year

OPTIONAL SLEEP STUDY ADD-ON Exclusion Criteria:

* Unable to undergo cardiac monitoring
* Unable to wear the sleep patch device for full monitoring period
* Implanted neurostimulator

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-08-15 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Emotional Ratings of Personal Memories (Memory Reconsolidation) | 2 days before and 1 day after treatment
  Negative/positive valence ratings associated with personal memories. A series of positive and negative adjectives will be presented to participants and they will have to rate on a scale of 1(not at all) to 10 (extremely) to what extent these words apply to how they feel when recalling the memory.

SECONDARY OUTCOMES:
Performance on Emotional Processing Tasks | Immediately before and after treatment and 1 day after treatment
  Performance on the Emotional Testing Battery (ETB), which contains an emotional word categorisation task, an emotional facial recognition task, and two emotional memory tasks.
Performance on Cognitive Flexibility Task | 1 day after treatment
  Performance on a probabilistic reversal learning task in which participants have to learn which strategy on a computer-task leads to a reward.
Performance on Response Inhibition Task | 1 day after treatment
  Performance on an emotional go/no-go task in which participants have to inhibit their responses to certain stimuli based on rules given at the start of each block of the task.

CONTACTS AND LOCATIONS:
Locations (1):
- Psychiatry Department, Oxford, United Kingdom